CLINICAL TRIAL: NCT01051167
Title: Bi-weekly Cetuximab Combined With FOLFOX-6 as First-line Treatment in Metastatic Colorectal Cancer Patients With Wild-type K-ras Status
Brief Title: Bi-weekly Cetuximab Combined With 5-fluorouracil/Leucovorin/Oxaliplatin (FOLFOX-6) in Metastatic Colorectal Cancer
Acronym: CEBIFOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Schuler, Prof. Dr. med. (Other)
Responsible Party: Sponsor-Investigator, Martin Schuler, Prof. Dr. med., Prof. Dr., Universität Duisburg-Essen
Organization: Universität Duisburg-Essen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT1-2007; 2007-000460-24 (EudraCT Number)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab + Folfox-6-regime (Experimental): Cetuximab 500 mg/m² administered as an intravenous infusion over 120 minutes on day 1 every 2 weeks. Combined with the following FOLFOX-6-regime:
  Oxaliplatin 85 mg/m² i.v. for 2 h on day 1, Folinic acid 400 mg/m² i.v. for 2 h concurrently with Oxaliplatin on day 1, Fluorouracil 400 mg/m² i.v. bolus after Folinic Acid on day 1, followed by Fluorouracil 2400 mg/m² i.v. over 46 h.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — 500 mg /m² cetuximab as an intravenous infusion over 120 minutes on day 1 every 2 weeks
  Other Names: Erbitux®

SUMMARY:
Cetuximab is normally given as a weekly schedule in the therapy of patients with metastatic colorectal cancer.

In order to improve the convenience for the patients in first line-therapy this study will evaluate the efficacy and safety of a bi-weekly combination of cetuximab with FOLFOX.

DETAILED DESCRIPTION:
For years the effective treatment of advanced colorectal carcinoma (CRC) was limited to fluorouracil (5-FU). Combination of 5-FU or a 5-FU analog with oxaliplatin, which has some antitumor activity as a single agent, shows synergistic activity. Combining oxaliplatin with a twice monthly folinic acid/5-FU schedule leads to a further improvement in first-line treatment of advanced CRC thus emerging to a standard regimen in first-line therapy of metastatic CRC.

Cetuximab is normally given as a weekly schedule. As recently shown a biweekly schedule with 500 mg/m² instead of the weekly standard regimen (initial dose of 400 mg/m² followed by 250 mg/m² every week) exhibits similar pharmacokinetic results with a comparable efficacy.

In order to improve the convenience for the patients, this study will evaluate the efficacy and safety of a bi-weekly combination of cetuximab with FOLFOX. Out of the various FOLFOX regimens the most convenient FOLFOX-6 schedule is chosen for the study, which has been tested before in two studies in combination with the standard weekly schedule of cetuximab. Recent data suggest a decreased efficacy of cetuximab in patients bearing a k-ras mutation in their CRC. Therefore only patients with no evidence for a mutated k-ras gene in the colorectal carcinoma cells will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic colorectal cancer
* Molecular test showing no mutation in the k-ras gene of colorectal carcinoma cells
* Male and female subjects ≥ 18 years of age
* 1st occurrence of metastatic disease (not curatively resectable)
* Life expectancy ≥ 12 weeks
* Presence of at least 1 bi-dimensionally measurable index lesion (not in an irradiated area)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at study entry
* Adequate bone marrow reserve:

leucocytes ≥ 3.0 x 109/l with neutrophils ≥ 1.5 x 109/l, platelets ≥ 100 x 109/l, haemoglobin ≥ 6.21 mmol/l (10 g/dl)

* Aspartate-aminotransferase (ASAT) and alanine-aminotransferase (ALAT) ≤ 2.5 x upper reference range, in case of liver metastasis ≤ 5 x upper reference range
* Serum creatinine ≤ 1.5 x upper reference range
* Bilirubin ≤ 1.5 x upper reference range
* Negative pregnancy test for female and effective contraception for both male and female subjects if the risk of conception exists
* Signed written informed consent

Exclusion Criteria:

* Evidence for a mutation of the k-ras gene in the colorectal carcinoma cells
* Previous exposure to epidermal growth factor receptor-targeting therapy
* Prior chemotherapy for metastatic disease
* Prior oxaliplatin based adjuvant chemotherapy or < 6 months after end of adjuvant treatment
* Other previous malignancy with exception of a history of a previous curatively treated basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Radiotherapy, surgery (excluding prior diagnostic biopsy) or any investigational drug in the 30 days before registration
* Concurrent chronic systemic immune therapy or hormone therapy not indicated in this study protocol
* Creatinine clearance < 30 ml/min
* Known hypersensitivity reaction to any of the components of study treatment
* Pregnancy (absence to be confirmed by ß-human chorionic gonadotropin (hCG) test) or lactation period
* Clinically relevant coronary artery disease, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Brain metastasis (known or suspected)
* Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
* Known alcohol or drug abuse
* Participation in another clinical study within the 30 days before registration
* Peripheral neuropathy > grade 1
* Significant disease which, in the investigator's opinion, would exclude the patient from the study
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Response rate (RECIST-Criteria) | Every 8 weeks

SECONDARY OUTCOMES:
Secondary objectives: Safety, Quality of life | Every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuler, Prof.Dr.med., Study Director — University of Duisburg-Essen Medical School
Locations (3):
- Germany (3):
  - University of Duisburg-Essen Medical School, Essen, North Rhine-Westphalia
  - Alfried Krupp von Bohlen und Halbach Krankenhaus gGmbH, Essen, North Rhine-Westphalia
  - Prosper Hospital Recklinghausen, Recklinghausen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasper S, Meiler J, Knipp H, Hohler T, Reimer P, Steinmetz T, Berger W, Linden G, Reis H, Markus P, Paul A, Dechene A, Schumacher B, Kostbade K, Virchow I, Ting S, Worm K, Schmid KW, Herold T, Wiesweg M, Schuler M, Trarbach T. Biweekly Cetuximab Plus FOLFOX6 as First-Line Therapy in Patients With RAS Wild-Type Metastatic Colorectal Cancer: The CEBIFOX Trial. Clin Colorectal Cancer. 2020 Dec;19(4):236-247.e6. doi: 10.1016/j.clcc.2020.03.003. Epub 2020 Mar 19. PMID 32737003